CLINICAL TRIAL: NCT03503357
Title: ConsCIOUS2: A Prospective Study of the Isolated Forearm Technique Commands, Long-term Sequelae and Electroencephalograph Correlates Following Laryngoscopy and Intubation in Patients 18 - 40 Years of Age
Brief Title: ConsCIOUS2 Study of the Isolated Forearm Technique Commands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Rambam Health Care Campus (Other); University of Groningen (Other); Centre Hospitalier Regional de la Citadelle (Unknown); RWTH Aachen University (Other); University of Pennsylvania (Other); Ludwig-Maximilians - University of Munich (Other); Cornell University (Other); Cairns Hospital (Unknown); Auckland District Health Board (Other Government); Waikato Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-0728; A530900 (Other: UW Madison); SMPH\ANESTHESIOLOGY\ANESTHESIO (Other: UW Madison)
Record Dates: First submitted 2018-03-27; First posted 2018-04-19 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia Awareness
Keywords: Consciousness; Electroencephalography; Anesthesia
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IFT Testing 1 (Experimental): Participants will be fitted with and IFT cuff and randomized to command list A intra-operatively to assess awareness.
  Interventions: Other: IFT Testing1
- IFT Testing 2 (Experimental): Participants will be fitted with and IFT cuff and randomized to command list B intra-operatively to assess awareness.
  Interventions: Other: IFT Testing 2
- IFT Testing 3 (Experimental): Participants will be fitted with and IFT cuff and randomized to command list C intra-operatively to assess awareness.
  Interventions: Other: IFT Testing 3
- IFT Testing 4 (Experimental): Participants will be fitted with and IFT cuff and randomized to command list D intra-operatively to assess awareness.
  Interventions: Other: IFT Testing 4

INTERVENTIONS:
Other: IFT Testing1 — Command List A
  Other Names: Command List A
  Arms: IFT Testing 1
Other: IFT Testing 2 — Command List B
  Other Names: Command List B
  Arms: IFT Testing 2
Other: IFT Testing 3 — Command List C
  Other Names: Command List C
  Arms: IFT Testing 3
Other: IFT Testing 4 — Command List D
  Other Names: Command List D
  Arms: IFT Testing 4

SUMMARY:
ConsCIOUS-2 is a multi-site study exploring the cognitive state of the Isolated Forearm Test (IFT) responder while under anesthetic.

DETAILED DESCRIPTION:
500 participants between the ages of 18-40 who will be undergoing surgery requiring general anesthetic will be recruited for this study. This study will use the Isolated Forearm Test (IFT) to identify patients at risk of anesthesia awareness. In the IFT, induction of anesthesia is followed by inflation of a cuff on the dominant arm before neuromuscular blockade (paralysis) is induced. The cuff prevents paralysis of the hand allowing the patient to communicate to an observer through predefined hand movements, typically following a command like: "Mrs. Jones, if you can hear me, squeeze my hand". Participants will thus be asked to follow a series of commands intraoperatively to assess awareness.

Routinely recorded clinical data will be collected to frame the observations about IFT responsiveness, and non-invasive EEG data will also be collected to provide information about the "brain state" of the patients. Patient reported confusion and objectively measured confusion using the Nurse Based Delirium Screening Tool (NuDesc) will be collected post operatively. Finally, participants will be contacted 24 hours and 7 days following their operation to complete an anesthesia satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years
2. English (or local language) competent
3. Informed consent obtained
4. Patients clinically requiring general anesthesia and intubation
5. Able to safely follow the IFT commands when awake and prior to their operation, per discretion of the PI.

Exclusion Criteria:

1. Age < 18 years old, >40 years old
2. Unable or unwilling to sign consent
3. Unable to undergo postoperative questions
4. Contraindication to IFT test such as unable to have tourniquet on arm for the IFT (e.g. lymphedema or operative site), rapid sequence inductions and requiring paralysis for laryngoscopy and intubation, per discretion of the PI.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Responsiveness | Intra-operative
  Identify the incidence of IFT responsiveness following intubation assessed by hand squeezing response following a randomized command sequence to assess for non-specific responses.

SECONDARY OUTCOMES:
Patient Reported Confusion Following Emergence | 15 minutes and 60 minutes after PACU admission
  Test the association between intra-operative IFT responsiveness and patient reported confusion following emergence from anesthesia and objectively assessed confusion using the NuDesc
EEG | Intra-operative
  Collect EEG data to identify monitoring patterns that discriminate responders and non-responders
Anesthesia Awareness with Recall | 24 hours and 7 days post-op
  Identify the incidence of implicit memory in post anesthesia care unit and anesthesia awareness with recall 24 hours and 7 days postoperatively using the structured Modified Brice questionnaire
Anesthesia Satisfaction | 24 hours and 7 days post-op
  Identify changes in patient satisfaction associated with IFT responsiveness via a patient satisfaction questionnaire administered 24 hours and 7 days postoperatively.
Predisposing Factors | Pre-operative
  Chart review of demographic factors that predispose to IFT responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sanders, MBBS, PhD, FRCA, Principal Investigator — University of Wisconsin, Madison
Locations (11):
- United States (3):
  - Cornell University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Cairns Hospital, Cairns, Australia
- Centre Hospitalier Regional de la Citadelle, Liège, Belgium
- Germany (2):
  - RWTH Aachen University, Aachen
  - University of Munich, Munich
- Rambam Health Care Campus, Haifa, Israel
- University of Groningen, Groningen, Netherlands
- New Zealand (2):
  - Auckland District Health Board, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No